CLINICAL TRIAL: NCT00175617
Title: Efficacy of Therapy With the Anti-androgen Spironolactone Compared to Topical Minoxidil in Female Pattern Hair Loss
Brief Title: Efficacy of Therapy With the Spironolactone Pills Compared to Minoxidil Lotion in Female Pattern Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05-0060
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Female Pattern Hair Loss
MeSH Terms: interventions — Spironolactone; Minoxidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Spironolactone — This study evaluates the efficacy of therapy with the anti-androgen spironolactone compared to topical minoxidil in female pattern hair loss.
Drug: Minoxidil — This study evaluates the efficacy of therapy with the anti-androgen spironolactone compared to topical minoxidil in female pattern hair loss.

SUMMARY:
This study evaluates the efficacy of therapy with the anti-androgen spironolactone compared to topical minoxidil in female pattern hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be premenopausal women older than 18 with female pattern hair loss.

Exclusion Criteria:

* Androgen excess
* Other scalp or hair disorders
* Contraindications to spironolactone treatment, especially pregnancy, electrolyte imbalances, history of breast cancer, or intake of interfering drugs
* Contraindications to minoxidil treatment, especially patients who are allergic to this treatment or have a history of low blood pressure or irregular heart beats

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-03-09 (Actual); Study Completion 2009-03-09 (Actual)

PRIMARY OUTCOMES:
hair density | after 3, 6 and 9 months

SECONDARY OUTCOMES:
percentage of subjects who experience side effects
subject assessment of treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Division of Dermatology, Hair Research and Treatment Centre, Vancouver, British Columbia, Canada